CLINICAL TRIAL: NCT04874974
Title: The PROBAS-Study: Developing a Process-based and Modular Group Therapy for Acute Psychiatric Patients With Psychotic Symptoms: a Single-arm Feasibility Study
Brief Title: Feasibility of a Novel Process-based Treatment for Patients With Psychosis
Acronym: PROBAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Max-Planck-Institute of Psychiatry (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-0025
Record Dates: First submitted 2021-04-26; First posted 2021-05-06 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Schizophrenia; Schizotypal Disorder; Delusional Disorder; Brief Psychotic Disorder; Shared Psychotic Disorder; Schizoaffective Disorder; Other Psychotic Disorder Not Due to A Substance or Known Physiological Condition; Unspecified Psychosis Not Due to a Substance or Known Physiological Condition; Manic Episode, Severe With Psychotic Symptoms; Bipolar Disorder, Current Episode Manic Severe With Psychotic Features; Bipolar Disorder, Current Episode Depressed, Severe, With Psychotic Features; Major Depressive Disorder, Single Episode, Severe With Psychotic Features; Major Depressive Disorder, Recurrent, Severe With Psychotic Symptoms
Keywords: Psychosis spectrum disorder; Process-based therapy; Modular psychotherapy; Group Therapy; Acceptance and Commitment Therapy (ACT); Metacognitive Training (MCT)
MeSH Terms: conditions — Schizophrenia; Schizotypal Personality Disorder; Schizophrenia, Paranoid; Psychotic Disorders; Shared Paranoid Disorder; Mania; Bipolar Disorder; Depressive Disorder, Major; Recurrence

STUDY DESIGN:
Intervention Model Description: Incoming patients from the clinic of Max Planck Institute of Psychiatry are continuously screened for study eligibility and - after they have given informed consent - are assigned to the experimental treatment condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Metacognitive and Defusion Training (Experimental): All participating patients are allocated to the same five-week experimental group therapy, which consists of three different modules (Module I: Psychoeducation on cognitive processes and rational of the therapy - week 1; Module II: Metacognition - week 2+3; Module III: Cognitive Defusion - week 4+5). Group therapy will start with a psychoeducation session of 60 minutes in the first week and will then take place twice a week with each session lasting 60 minutes.
  Interventions: Behavioral: Metacognitive and Defusion Training

INTERVENTIONS:
Behavioral: Metacognitive and Defusion Training — Module I will give a brief introduction into the rational of the therapy and explain the terms cognitive biases and relational responding and their role in the development of psychological problems (psychosis) in a simple language and with the help of examples and small exercises. The principle of metacognition and cognitive defusion in psychotherapy will be made clear. An outlook on the procedures and the goals of the group therapy will be given. Module II will include interventions adapted from the MCT manual (Moritz et al., 2017) and Module III with consist of defusion strategies taken from the ACT group manual (Dambacher et al., 2020) and existing studies on ACT and psychosis (Bach et al., 2013; Gaudiano & Herbert, 2006).

SUMMARY:
The purpose of this single-arm feasibility study is to develop and pilot test a novel process-based and modular group therapy approach for patients with acute psychotic symptoms in an inpatient setting.

DETAILED DESCRIPTION:
Due to the enormous economic and social costs of psychotic-spectrum disorders, increasing the effectiveness of treatment options has become an important subject for psychiatric research. Latest findings in the field of psychotherapy for psychosis show some promising results for so-called Process-based Therapies (PBT) such as the Metacognitive Training (MCT) and Acceptance and Commitment Therapy (ACT) (Barnicot et al., 2020). Instead of trying to change the content of psychotic symptoms such as hallucinations and delusions, PBT directly address cognitive processes, which have been found to maintain the disorder's symptomatology (Hayes et al., 2020). While MCT focusses on changing patients' cognitive biases by inducing metacognition (Moritz & Woodward, 2007), ACT works with psychological processes such as mindfulness, willingness and cognitive distancing (Gaudiano & Herbert, 2006). There is a growing study base for PBT in a psychotic outpatient setting, research in non-ambulatory settings though is rare (Barnicot et al., 2020). Therefore, the aim of the current study is to develop and test the feasibility and safety of a new process-based group therapy program for acute psychotic patients. The five-week treatment approach will consist of three different modules combining interventions from both MCT and ACT (Module I: Psychoeducation, Module II: Metacognition, Module III: Cognitive Defusion). First preliminary effectiveness and process measures (PANSS, BPRS, WHO-DAS, CGI, BCIS and CFQ) will also be included in order to inform the design of future research. Thus, the study will give valuables insights in the feasibility and effectiveness of an innovative psychotherapy approach and breaks new ground in the field of psychotherapy research for psychosis.

ELIGIBILITY:
Inclusion Criteria:

* Main diagnosis of a mental disorder with psychotic symptoms according to ICD-10 criteria currently experiencing delusions and hallucinations (F20, F21, F22, F23, F24, F25, F28, F29, F30.2, F31.2, F31.5, F32.3, F33.3) indicated by diagnostic assessment of attending MD
* Age between 18 and 70 years
* Informed consent to the study procedures and assessments (in written form)

Exclusion Criteria:

* Severe neurological or internal concomitant diseases
* IQ < 80; severe learning disability, brain damage or pervasive developmental disorder
* Missing eligibility for psychotherapy because of missing language skills/hostile or uncooperative behaviour.

No further constraints will be imposed in order to collect data in a representative clinical sample.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2023-09-23 (Actual)

PRIMARY OUTCOMES:
Eligibility rate | assessed from study start in May 2021 until study completition in May 2022, up to 1 year
  proportion of those eligible to participate as a percentage of those screened
Consent rate | assessed from study start in May 2021 until study completition in May 2022, up to 1 year
  proportion of those who signed the informed consent as a percentage of those who where approached to participate
Trial entry rate | assessed from study start in May 2021 until study completition in May 2022, up to 1 year
  proportion of those who consented and completed baseline measures
Completion rate | assessed from study start in May 2021 until study completition in May 2022, up to 1 year
  proportion of assessments completed at each time point including screening, baseline, intervention and final meeting and reasons for missing data; subjective patient feedback on frequency, duration, delivery, method and content of the assesments
Missing data rate | assessed from study start in May 2021 until study completition in May 2022, up to 1 year
  proportion of missing data for each time point including screening, baseline, intervention and final meeting
Patient engagement | assessed from study start in May 2021 until study completition in May 2022, up to 1 year
  frequency of unattended sessions per patient as well as the reason for non-attendance
Drop out rate | assessed from study start in May 2021 until study completition in May 2022, up to 1 year
  proportion of patients who entered the trial, attended at least one therapy session after baseline but decided to drop out as well as reasons for the drop out
Adverse events | assessed from study start in May 2021 until study completition in May 2022, up to 1 year
  number and nature of adverse events
Acceptability of Module I | after completion of Module I in week 1
  self-rating on subjective effectiveness and acceptability of Module I (one session Psychoeducation). The questionnaire will be designed in a manner similar to session feedback forms developed by Moritz and Woodward (2007) including likert-scaled items on satisfaction, effectiveness, usefulness, applicability and transparency of the aim as well as open-ended feedback
Acceptability of Module II | after completion of Module II in week 3
  self-rating on subjective effectiveness and acceptability of Module II (four sessions Metacognition). The questionnaire will be designed in a manner similar to session feedback forms developed by Moritz and Woodward (2007) including likert-scaled items on satisfaction, effectiveness, usefulness, applicability and transparency of the aim as well as open-ended feedback
Acceptability of Module III | after completion of Module III in week 5
  self-rating on subjective effectiveness and acceptability of Module III (four sessions Cognitive Defusion). The questionnaire will be designed in a manner similar to session feedback forms developed by Moritz and Woodward (2007) including likert-scaled items on satisfaction, effectiveness, usefulness, applicability and transparency of the aim as well as open-ended feedback
Semi-structured interviews | after completing Module III in week 5
  conducted with one randomly selected patient out of every therapy cycle after completion; selected patients will be asked in detail about feasibility and perceived efficacy of the group program

SECONDARY OUTCOMES:
Psychopathological in general and positive and negative psychotic symptoms (PANSS) | before session 1 in week 1 and after completing the therapy in week 5
  assessed with the semi-structured clinical interview Positive and Negative Syndrome Scale (PANSS), the internationally most widely used measure of psychotic symptomatology. The scale ranges from a minimum of 30 (no symptomatology) up to a maximum of 126 (severe symptomatology)
Psychopathological in general and positive and negative psychotic symptoms (BPRS) | before session 1 in week 1 and after completing the therapy in week 5
  assessed with the semi-structured clinical interview Brief Psychiatric rating scale (BPRS), next to PANSS the internationally second most used measure of psychotic symptomatology. The scale ranges from a minimum of 18 (no symptomatology) up to 210 (severe symptomatology)
Positive symptoms (hallucinatiosn and delusions) and their severity, intensity and frequency (PSYRATS) | before session 1 in week 1 and after completing the therapy in week 5
  measured with the clinical interview Psychotic Symptom Rating Scale (PSYRATS). The subscale auditory hallucinations ranges from a minimum of 0 (no distress) up to a maximum of 44 (high distress), the subscale delusions from a minimum of 0 (no distress) up to a maximum of 24 (high distress)
Patient's improvement (CGI) | The patient's supervising MD will rate CGI's severity scale for each patient in week 1 and week 5, and the improvement scale only after week 5
  will be gathered with the Clinical Global Impression Scale (CGI). The Severity scale ranges from a minimum of 1 (not at all ill) up to a maximum of 7 (among the most ill patients) and the Improvement scale from a minimum of 1 (very much improved) up to a maximum of 7 (very much worse)
Social functioning (WHODAS) | in week 1 and week 5
  social functioning will be self-administered by patients through the World Health Organisation Disability Assessment Schedule (WHODAS).
Therapy processes of metacognition (BCIS) | before starting Module II in week 2 and after completing Module II in week 3
  Beck's Cognitive Insight Scale (BCIS) will be filled in from patients to measure cognitive insight. Scores on the subscale Self-reflectiveness range from a minimum of 0 (high self-reflectiveness) to a maximum of 36 (high self-reflectiveness), scores on the subscale Self-Certainty range from a minimum of 0 (high self-certainty) to a maximum of 24 (low self-certainty)
Degree of Cognitive fusion (CFQ) | before starting Module III in week 4 and after completing Module II in week 5
  The Cognitive Fusion Questionnaire (CFQ) will be surveyed from patients to measure the degree of cognitive fusion. The scale ranges from a minimum of 7 (low cognitive fusion) up to a maximum of 49 (high cognitive fusion)

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Lucae, MD, Prof., Principal Investigator — Max-Planck-Institute of Psychiatry; Johannes M Kopf-Beck, PhD, Principal Investigator — Max-Planck-Institute of Psychiatry
Locations (1):
- Max Planck Institute of Psychiatry, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barnicot K, Michael C, Trione E, Lang S, Saunders T, Sharp M, Crawford MJ. Psychological interventions for acute psychiatric inpatients with schizophrenia-spectrum disorders: A systematic review and meta-analysis. Clin Psychol Rev. 2020 Dec;82:101929. doi: 10.1016/j.cpr.2020.101929. Epub 2020 Oct 17. PMID 33126038
- [Background] Moritz S, Woodward TS. Metacognitive training in schizophrenia: from basic research to knowledge translation and intervention. Curr Opin Psychiatry. 2007 Nov;20(6):619-25. doi: 10.1097/YCO.0b013e3282f0b8ed. PMID 17921766
- [Background] Gaudiano BA, Herbert JD. Acute treatment of inpatients with psychotic symptoms using Acceptance and Commitment Therapy: pilot results. Behav Res Ther. 2006 Mar;44(3):415-37. doi: 10.1016/j.brat.2005.02.007. PMID 15893293
- [Background] Hayes SC, Hofmann SG, Ciarrochi J. A process-based approach to psychological diagnosis and treatment:The conceptual and treatment utility of an extended evolutionary meta model. Clin Psychol Rev. 2020 Dec;82:101908. doi: 10.1016/j.cpr.2020.101908. Epub 2020 Sep 7. PMID 32932093